CLINICAL TRIAL: NCT06954532
Title: ADIE-BC - Aligning Dimensions of Interoceptive Experience in Breast Cancer Survivors
Acronym: ADIE-BC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University College, London (Other); Brighton & Sussex Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR/DP-23/24-41430
Record Dates: First submitted 2025-04-09; First posted 2025-05-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Primary Breast Cancer
Keywords: Breast Cancer; Primary Breast Cancer; ADIE Therapy; Biobehavioral Medicine; Anxiety Management; Interoception; Emotion Regulation; Interoceptive Training; Cardiac Interoception; Mind-Body Therapy
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: This is an open-label, single arm pilot study, in which all participants will receive ADIE Therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADIE Therapy (Experimental): Participants will undergo 6 sessions of cardiac interoceptive training (ADIE Therapy).
  Interventions: Behavioral: Interoceptive training

INTERVENTIONS:
Behavioral: Interoceptive training — There will be 6 interoceptive training sessions. Each training session will comprise two blocks, between which participants will undergo a self-paced, light physical activity that aims to enhance heartbeat perception and lasts 2 to 3 minutes. During the pre- and post-exercise block, each participant will complete cardiac interoceptive tasks, and for each trial, note their confidence in their answer on a visual analogue scale and then be given accurate feedback about their objective heartbeat perception accuracy, relative to their objective accuracy.

SUMMARY:
A breast cancer diagnosis can lead to significant anxiety, and for many survivors, this anxiety continues well beyond the end of treatment. While standard anxiety therapies are helpful for some, these therapies often fall short for breast cancer survivors due to an individual's unique experience-particularly changes in how survivors perceive and relate to the body, a process known as interoception.

The study will evaluate the feasibility and acceptability of a novel interoceptive training approach called ADIE Therapy. ADIE Therapy trains participants to better recognise bodily signals, and has shown promising results in reducing anxiety in non-cancer populations. The aim of the study is to assess the acceptability and feasibility of ADIE Therapy for breast cancer survivors.

DETAILED DESCRIPTION:
Anxiety is a common and often long-lasting psychological consequence of a breast cancer diagnosis. Post-cancer anxiety frequently co-occurs with somatic symptoms such as persistent pain and fatigue. For many individuals, feelings of anxiety do not resolve with the completion of cancer treatment and can persist for months or even years. For yet others, anxiety increases after cancer treatment has ended. Although standard therapies-such as cognitive behavioural therapy or pharmacological interventions-can be effective for some, these interventions do not adequately address the needs of all breast cancer survivors. This may be due, in part, to the unique physical and emotional challenges faced by this group, including changes in the way internal bodily sensations are experienced and interpreted.

Interoception refers to the process by which the nervous system senses, interprets and integrates information from inside the body. ADIE Therapy - which stands for Aligning Dimensions of Interoceptive Experience - has shown promise as a novel interoceptive intervention to reduce anxiety and somatic symptoms in non-cancer populations. ADIE Therapy uses simple, biofeedback-based tasks to enhance precision in perceiving cardiac interoceptive signals.

The primary aim of the study is to demonstrate the acceptability and feasibility of ADIE Therapy for survivors of primary breast cancer. A mixed-methods approach will be used to evaluate the feasibility and acceptability of ADIE Therapy, incorporating both quantitative and qualitative measures. Secondary aims include ascertaining whether ADIE Therapy leads to improvements in interoceptive measurements (including self-reported interoceptive sensibility and objective interoceptive markers), anxiety symptoms (including generalised and cancer-specific anxiety), depressive symptoms, somatic symptoms, and body mindsets. Additional secondary aims include exploring the feasibility of incorporating blood and saliva collection into the ADIE-BC research protocol, which could facilitate assessment of biomarker outcomes in a future randomised controlled trial of ADIE-BC.

Participants will be recruited through charity and foundation partners, as well as through community settings. ADIE Therapy involves the administration of simple biofeedback-based tasks designed to progressively improve objective interoceptive accuracy, specifically through cardiac interoceptive exercises. A schedule of six interoceptive training sessions will be agreed with each participant, with the option to complete intermediate training sessions either in-person or at home. During each training session, participants will complete the cardiac interoceptive tasks with active feedback, before and after a 2-to-3-minute period of self-directed exercise, intended to elevate heart rate. The resulting cardiovascular arousal aims to amplify sensations associated with the heartbeat, thereby facilitating perception during interoceptive tasks. In addition to training, participants will complete three interoceptive assessments conducted at pre-training, midpoint (Week 4), and post-training (Week 7), each scheduled within a ±2-week window. A series of questionnaires will also be administered before and after training. All participants will complete a semi-structured exit interview to provide feedback on their experience of participating in ADIE Therapy. Participants who complete the study will be invited to take part in an optional three-month follow-up assessment (Week 18), which repeats the same interoceptive tasks and questionnaires to evaluate longer-term effects of the therapy.

The present study is an open-label, single-arm acceptability and feasibility study. The investigators aim to recruit a total of 20 participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Residing in the UK and able to travel into London
* Can read and write in English
* Have had a diagnosis of Primary Breast Cancer
* Have completed active, hospital-based treatment for primary breast cancer (Stages 1, 2 or 3; this refers to radiotherapy, surgery, or chemotherapy) 6 months - 10 years previously (this does not apply to ongoing endocrine (hormone) therapy)

Exclusion Criteria:

* Currently taking medication for cardiac arrhythmia (e.g., beta blockers)
* Currently in active treatment for breast cancer and/or other types of cancer
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the Intervention - Theoretical Framework of Acceptability (TFA) Questionnaire | Post-Treatment (Week 7)
  Acceptability will be assessed quantitatively at the end of treatment through a brief survey related to acceptability, including ease of use, satisfaction, and overall experience. Survey responses will be reported categorically. Responses are measured using a five-point Likert scale from 'Strongly disagree' to 'Strongly agree' with higher scores indicating greater acceptability.
Feasibility and Acceptability of the Intervention - Qualitative Interview | Post-Treatment (Week 7)
  Feasibility and acceptability will be assessed at the end of treatment through semi-structured interviews exploring participants' experiences with the intervention, including ease of use, comprehensibility, perceived usefulness, barriers to participation, and suggestions for improvement. Qualitative responses will be described and summarized.
Acceptability of the Intervention - Net Promoter Score | Post-Treatment (Week 7)
  Acceptability will be evaluated by examining mean promoter score (measured on 10-point Likert scale) post intervention. Range 0-10 (higher scores indicate more acceptability).
Feasibility of the Study - Participant Retention | Baseline through Post-Treatment (Week 7)
  Retention rates will be assessed by tracking the proportion of participants who complete the full ADIE Therapy programme, including all scheduled training sessions and study assessments.
Feasibility of the Study - Session Adherence | Baseline through Post-Treatment (Week 7)
  Session adherence will be assessed by tracking attendance across the six scheduled interoceptive training sessions. Adherence will be calculated as the proportion of completed sessions per participant.

SECONDARY OUTCOMES:
Cardiac Interoceptive Accuracy, Awareness, and Sensibility Scores | Baseline, Midpoint (Week 4), Post-Treatment (Week 7), and 3-month Follow-Up (Week 18; optional)
  Interoceptive outcomes will be assessed using heartbeat detection tasks to evaluate three domains of cardiac interoception:
  1. Accuracy (objective performance on heartbeat detection tasks)
  2. Sensibility (subjective confidence or perception of performance)
  3. Awareness (metacognitive insight into accuracy, i.e., the correspondence between confidence and actual performance).
  These measures will be collected to assess participants' interoceptive processing during the intervention.
Generalized Anxiety Disorder (GAD-7) | Baseline, Midpoint (Week 4), Post-Treatment (Week 7), and 3-month Follow-Up (Week 18; optional)
  The GAD-7 assesses core symptoms and signs of anxiety with 7 items. Participants respond on a four-point scale based on their experience of anxiety over the past two weeks.
Spielberger State-Trait Anxiety Inventory (STAI) | Baseline, Midpoint (Week 4), Post-Treatment (Week 7), and 3-month Follow-Up (Week 18; optional)
  The STAI assesses both state anxiety (temporary) and trait anxiety (general tendency) with 40 items, 20 for state anxiety and 20 for trait anxiety. Items are rated on a four-point scale.
Patient Health Questionnaire (PHQ-8) | Baseline, Midpoint (Week 4), Post-Treatment (Week 7), and 3-month Follow-Up (Week 18; optional)
  The PHQ-8 measures core symptoms and signs of depression. Participants respond on a four-point scale based on their experience over the last two weeks.
Anxiety Sensitivity Index (ASI) | Baseline, Midpoint (Week 4), Post-Treatment (Week 7), and 3-month Follow-Up (Week 18; optional)
  The ASI evaluates concerns about anxiety and its potential consequences. The ASI is comprised of 16 items rated on a four-point scale.
Toronto Alexithymia Scale (TAS-20) | Baseline, Midpoint (Week 4), Post-Treatment (Week 7), and 3-month Follow-Up (Week 18; optional)
  The TAS-20 assesses difficulty in identifying and describing emotions. The TAS-20 consists of 20 items rated on a four-point scale.
Fear of Cancer Recurrence Inventory - Short Form (FCRI-SF) | Baseline, Midpoint (Week 4), Post-Treatment (Week 7), and 3-month Follow-Up (Week 18; optional)
  The FCRI-SF assesses participants' fears of cancer recurrence and how this impacts their lives. It consists of 9 items, with a mix of five-point scales and specific frequency/perceived risk questions.
Body Perceptions Questionnaire (BPQ) - Body Awareness Short Form | Baseline, Midpoint (Week 4), Post-Treatment (Week 7), and 3-month Follow-Up (Week 18; optional)
  A measure of sensitivity for internal bodily functions with 26 items. Values at the high end of the scale reflect hypersensitivity and values at the low scale reflect hyposensitivity.
Multidimensional Assessment of Interoceptive Awareness (MAIA-2) | Baseline, Midpoint (Week 4), Post-Treatment (Week 7), and 3-month Follow-Up (Week 18; optional)
  The MAIA-2 assesses various dimensions of interoception with 37 items. It contains 8 subscales assessing 5 dimensions of body awareness.
Bodily Threat Monitoring Scale (BTMS) | Baseline, Midpoint (Week 4), Post-Treatment (Week 7), and 3-month Follow-Up (Week 18; optional)
  Bodily threat monitoring will be assessed via a 19-item self-report measure, rated on a five-point scale. Higher scores indicate greater propensity to monitor the body for threatening signs and symptoms.
Body Mindset Inventory - Version 2 (BMI-2) | Baseline, Midpoint (Week 4), Post-Treatment (Week 7), and 3-month Follow-Up (Week 18; optional)
  The BMI-2 assesses mindsets participants may hold about their body in the context of chronic disease. Participants respond by indicating how much they agree with each statement on a six-point scale.
EuroQoL 5 Dimensions, 5 Levels (EQ-5D-5L) | Baseline, Midpoint (Week 4), Post-Treatment (Week 7), and 3-month Follow-Up (Week 18; optional)
  The EQ-5D-5L measures five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression).
Pain Intensity, Interference, and Body Location | Baseline, Midpoint (Week 4), Post-Treatment (Week 7), and 3-month Follow-Up (Week 18; optional)
  The PROMIS interference and intensity measures, as well as items from the Graded Chronic Pain Scale-Revised (Von Korff et al., 2020) and the body map from the Brief Pain Inventory (Cleeland et al, 1994) will be used to assess pain.
Patient Global Impression of Change (PGIC) Scale | Post-Treatment (Week 7)
  Single question asking participants to rate how their condition has changed since a specified point in time, with lower scores indicating greater degree of improvement.

OTHER OUTCOMES:
Salivary and Blood-Based Biomarkers | Assessed at Baseline and Post-Treatment (Week 7)
  Saliva and blood samples will be collected pre-treatment and post-treatment (Week 7) to explore the feasibility of incorporating biomarker collection into the ADIE-BC research protocol.
Adverse Events Monitoring | Structured questions Post-Treatment (Week 7); Open-text form available continuously throughout participation.
  Adverse events will be monitored using a protocol adapted from Wileman et al. (2024) for digital trials. Participants will complete structured questions assessing physical, psychological, or other adverse events at post-treatment (Week 7). An open-text form will also be available throughout the study, allowing participants to report any adverse experiences at any time.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren C. Heathcote, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be shared with other researchers to comply with open science practices.
Time Frame: De-identified IPD will be shared on an online, open science data repository platform from the time that the study has been published and will be available indefinitely.
Access Criteria: De-identified IPD will be available open access.

REFERENCES:
- [Background] Quadt L, Garfinkel SN, Mulcahy JS, Larsson DE, Silva M, Jones AM, Strauss C, Critchley HD. Interoceptive training to target anxiety in autistic adults (ADIE): A single-center, superiority randomized controlled trial. EClinicalMedicine. 2021 Aug 1;39:101042. doi: 10.1016/j.eclinm.2021.101042. eCollection 2021 Sep. PMID 34401684